CLINICAL TRIAL: NCT01177579
Title: Human Biomarkers for Assessing Copper Deficiency and Repletion: A Pilot Study
Brief Title: Human Biomarkers for Assessing Copper Deficiency
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Nana Gletsu-Miller, Assistant Professor, Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 00006969
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Copper Deficiency
Keywords: Bariatric surgery, copper deficiency, biomarkers
MeSH Terms: interventions — Gluconates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aim 1; Biomarkers (No Intervention): Blood concentrations of copper coenzymes will be monitored for 1 year
- Copper supplement Arm (Experimental): 4 mg or 8 mg copper will be compared in a randomized controlled study
  Interventions: Dietary Supplement: Copper gluconate
- Normal Controls (No Intervention): Normal subjects will be used to generate reference measures.

INTERVENTIONS:
Dietary Supplement: Copper gluconate — 4 or 8 mg copper gluconate/day will be assessed for efficacy of copper repletion
  Arms: Copper supplement Arm

SUMMARY:
Copper is an essential nutrient for humans and is cofactor in enzymes that participate in critical body functions. Insufficient copper can lead to hematological and neurological abnormalities that may be irreversible if left untreated. Copper deficiency is believed to be rare in the U.S. population because typical dietary intake is usually sufficient to meet requirements. More recent evidence suggests that specific populations may be susceptible to copper deficiency in cases where copper absorption in the gut is impaired following gastric surgery or in individuals with high intakes of zinc. Preliminary studies by us and others have identified significant levels of moderate and severe symptomatic copper deficiency in patients who have undergone weight loss (bariatric) gastric bypass surgery. Copper deficiency in humans is difficult to recognize and treat because current diagnostic tools rely on measures of plasma concentrations of copper and ceruloplasmin, which are neither sensitive nor specific for copper deficiency, and early warning blood markers (biomarkers) have not been identified. Recent developments indicate that copper chaperone molecules and cuproenzymes such as cytochrome C oxidase and superoxide dismutase may be more sensitive to changes in copper status, but there has been very little work done in humans. The studies outlined here are aimed at assessing copper status using these biomarkers in gastric bypass surgery patients who are at risk for symptomatic copper deficiency. In addition, patients identified to be deficient will be supplemented with copper and this treatment will be evaluated using biomarker concentrations. The findings of these studies should provide insight into the effectiveness of novel biomarkers to identify those at risk and to guide appropriate treatment to prevent serious and permanent morbidity due to copper deficiency.

ELIGIBILITY:
CuD subjects In order to be enrolled into the CuD Arm, subjects who have had RYGB surgery will be recruited and screened for eligibility (inclusion and exclusion criteria below). Subjects whose plasma copper concentrations are in the deficient range (less than 80 μg/dL for women and less than 70 µg/dL for men, and/or ceruloplasmin activity below 62 units/L-1) following 4 weeks of supplementation with the RDA for copper will be eligible. Such supplementation is the routine standard of care with all patients undergoing RYGB surgery. This process aims to exclude patients who were only marginally copper deficient and not in need of sustained copper therapy. Subjects will be notified about their copper status by a study physician. They will be contacted by the study team, and their willingness to participate in the study will be determined.

Inclusion criteria: 1) Patient has a history of RYGB weight loss surgery; 2) subject has a plasma copper level which is less than 80 μg/dL for women andl less than 70 µg/dL for men, and/or ceruloplasmin activity below 62 units/L-1; 3) subject is at least 18 but not more than 65 years of age; and 4) subject has signed an informed consent.

Exclusion criteria: 1) subject exhibits severe neurologic signs or symptoms (e.g. severe paresthesias, severe gait disturbances, or severe weakness which require intravenous copper supplementation; 2) subject is pregnant; 3) subject has history of surgical revision or conversion of bariatric procedure; 4) subject has a history of hospitalization for acute illness in the previous 3 months; 5) subject has current active malignant neoplasm; or history of malignancy other than localized basal cell cancer of skin during previous 5 years; 6) subject has current history of type 1 or type 2 diabetes mellitus.

CuN subjects In order to be enrolled into the CuN control arm, subjects who have had RYGB surgery will be recruited and screened for eligibility (inclusion and exclusion criteria below). Subjects will have plasma copper concentrations in the normal range (80 - 155 μg/dL for women and 70 - 140 µg/dL for men, and/or ceruloplasmin activity above 62 units/L-1). Subjects will also be eligible if they can be matched for stage of weight management (either active weight loss or weight stable) and gender with a CuD subject. Subjects will be notified about their copper status and their eligibility and their willingness to participate in the study will be determined.

Inclusion criteria: 1) Patient has a history of RYGB weight loss surgery; 2) subject has a plasma copper level which is 80 - 155 μg/dL for women and 70 - 140 µg/dL for men, and/or ceruloplasmin activity above 62 units/L-1; 3) subject can be matched for stage of weight management and gender with a CuD subject, 4) subject is at least 18 but not more than 65 years of age; and 5) subject has signed an informed consent.

Exclusion criteria: 1) subject is pregnant; 2) subject has history of surgical revision or conversion of bariatric procedure; 3) subject has a history of hospitalization for acute illness in the previous 3 months; 4) subject has current active malignant neoplasm; or history of malignancy other than localized basal cell cancer of skin during previous 5 years; 5) subject has current history type 1 or type 2 diabetes mellitus.

NW Control Arm For the normal-weight control arm (NW Control), subjects who have not had bariatric surgery and are of normal weight will be recruited.

Inclusion criteria: 1) Subject has a plasma copper level which is 80 - 155 μg/dL for women and 70 - 140 µg/dL for men, and/or ceruloplasmin activity above 62 units/L-1; 2) subject is of normal weight, BMI between 20 - 30 kg/m2, 3) subject is at least 18 but not more than 65 years of age; and 4) subject has signed an informed consent.

Exclusion criteria: 1) subject is pregnant; 2) subject has history of abdominal surgery or history of gastrointestinal disease; 3) subject has a history of hospitalization for acute illness in the previous 3 months; 4) subject has current active malignant neoplasm; or history of malignancy other than localized basal cell cancer of skin during previous 5 years; 5) subject has current history type 1 or type 2 diabetes mellitus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-11; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
copper co-enzymes | 1 year
  expression of CCS, SOD and COX4 in blood samples

SECONDARY OUTCOMES:
blood copper concentrations | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States